CLINICAL TRIAL: NCT03459482
Title: Endpoint Determination Study for An Antibody Guided Dietary Restriction Trial Using Biomerica InFoods® IBS Test in Patients With a Previous Diagnosis of Irritable Bowel Syndrome (IBS)
Brief Title: Endpoint Determination Study Protocol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biomerica (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EPT-InF24-001
Record Dates: First submitted 2018-02-20; First posted 2018-03-09 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-08

CONDITIONS: Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Intervention Model Description: Parallel Design
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 - True Food Elimination Diet (Experimental): Group 1 (experimental group): Subjects will be given an elimination diet based upon foods with a positive antibody profile in the Biomerica InFoods® IBS test. The elimination diet will also exclude any and all foods to which the subject has a known IgE allergy and foods the subject already currently eliminates.
  Interventions: Other: Food Elimination Diet
- Group 2 - Sham Food Elimination Diet (Sham Comparator): Group 2 (control group): Subjects will be given a "Sham" elimination diet. The sham diet will eliminate the same number of foods but none of the actual foods to which the patient had a positive antibody profile in the Biomerica InFoods® IBS test. The sham diet will also eliminate any and all foods to which the subject has a known IgE allergy and foods the subject already currently eliminates.
  Interventions: Other: Food Elimination Diet

INTERVENTIONS:
Other: Food Elimination Diet — Subjects asked to participate in a food elimination diet, either True or Sham to evaluate the effects on their IBS symptoms

SUMMARY:
This study is designed to evaluate the most applicable endpoints for evaluation of the Biomerica InFoods® IBS product.

DETAILED DESCRIPTION:
The objective of this Endpoint Determination Study is to address key elements regarding a proposed larger clinical study design:

1. Comparing different potential primary outcome measures
2. Demonstrating that an exclusionary diet as determined by elevated IgG levels using the Biomerica InFoods® IBS Test is associated with alleviation of IBS symptoms
3. Demonstrating the ability to mask the sham diet
4. Demonstrating the safety of the exclusionary diet

Subjects' diets will be based on the results of the Biomerica, InFoods® IBS Test.

Immunoglobulin G (IgG) levels above a certain threshold are considered a positive response against a specific food or foods. It is expected that severity of symptoms of IBS will decrease when foods that generate a positive immune response in the Biomerica InFoods® IBS test are eliminated from the diet of the IBS patient.

The Endpoint Determination Study format will be a double-blinded randomized controlled clinical study enrolling subjects at two trial sites within the United States and designed to evaluate the use of IgG antibody guided dietary restrictions, based on the Biomerica InFoods® IBS Test, in the management of patients diagnosed with Irritable Bowel Syndrome (IBS).

The 2 sites will enroll approximately equal numbers of subjects. The target for each site is a minimum of 30 subjects in each classification: IBS with diarrhea [IBS-D], IBS with constipation [IBS-C] and IBS mixed [IBS-M] for a minimum of 90 patients per site, 180 total subjects for this study.

ELIGIBILITY:
Inclusion Criteria:

* 21 years old or older.
* Able to read and understand English.
* Willing and able to sign the informed consent.
* Have access to a computer and/or cell phone access for Electronic Data Capture (EDC)
* Meets Rome IV Diagnostic Criteria for IBS
* Willing to follow a food elimination die
* Well controlled diabetic patients; A1C <7.5 and stable medication (>3 months, NOT Metformin
* Score between ≥ 3 and <7.5 on the Abdominal Pain Intensity Assessment (IBS_API) based on a weekly average of worst daily (in past 24 hours) abdominal pain on a 0 to 10 point scale.
* Patients who are on stable (> 3 months) doses of medications or treatments for their IBS (e.g., probiotics, fiber, Viberzi, Linzess, Amitiza, Alosetron, Plecanatide, anticholinergics, antidepressants, Zofran bile acid sequestrants, or anti-diarrheals) will be allowed to continue their medications as long as no change in treatment is planned for the duration of the study and no dose adjustment is made during the duration of the study.
* A positive IgG antibody response for at least one food in the Biomerica InFoods® IBS panel

Exclusion Criteria:

* Unable to provide consent.
* Cannot use EDC system due to no cell phone and no computer access
* Does not qualify for a diagnosis of IBS by IV Diagnostic Criteria
* Diagnosed IBS, but an IBS-API score of <3.0 and >7.5
* Pregnant or breastfeeding
* Patients with diabetes currently on Metformin
* Patients who have used Rifaximin in the past 3 months
* Patients engaged in another type of diet therapy, i.e. FODMAP
* Patients which physicians are anticipating starting a new medication, change in dosage, diet or other treatment for IBS during the study
* Chronic pain from other conditions besides IBS
* Current or previous use of narcotic medications within past 3 months
* History of prior GI surgery except for cholecystectomy or appendectomy.
* History with any of the following:

Gastroparesis, Uncontrolled GERD, Anorexia/bulimia Celiac disease Crohn's disease, Ulcerative Colitis, Abdominal/gastro cancer(s), Malabsorption syndrome(s).

* History of any other relevant inter-current medical conditions that could interfere with their participation in the study or the objectives of the study
* History of psychosis, schizophrenia, mania, or major psychiatric illness needing hospitalization within the past 6 months

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 556 (Actual)
Dates: Start 2018-06-21 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Change in the IBS-API - Abdominal Pain Intensity. The IBS-API is being assessed daily from enrollment (baseline) to study completion; total 10 weeks | Daily for 10 weeks
  Abdominal pain intensity will be measured daily using an 11-point (0-10) numeric rating scale (NRS) that asks subjects to rate their worst abdominal pain over the past 24-hours.

CONTACTS AND LOCATIONS:
Overall Officials: William D Chey, MD, Principal Investigator — University of Michigan; Anthony J Lembo, MD, Principal Investigator — Beth Israel Deaconess Medical Center (Harvard)
Locations (8):
- United States (8):
  - Mayo Clinic, Scottsdale, Arizona
  - Mayo Clinic, Jacksonville, Florida
  - Family Medicine Specialists, Wauconda, Illinois
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Michigan Health System, Ann Arbor, Michigan
  - Houston Methodist Research Institute, Houston, Texas
  - UT Health, Houston, Texas
  - Gastroenterology Research of San Antonio, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No
It is not yet known if there will be a plan to make IPD available.

REFERENCES:
- [Derived] Singh P, Chey WD, Takakura W, Cash BD, Lacy BE, Quigley EMM, Randall CW, Lembo A. A Novel, IBS-Specific IgG ELISA-Based Elimination Diet in Irritable Bowel Syndrome: A Randomized, Sham-Controlled Trial. Gastroenterology. 2025 Jun;168(6):1128-1136.e4. doi: 10.1053/j.gastro.2025.01.223. Epub 2025 Jan 31. PMID 39894284